CLINICAL TRIAL: NCT03729895
Title: Clinical Effect and Upper Airway Changes of Customized Adjustable Oral Appliance in the Treatment of Patients With Obstructive Sleep Apnea Syndrome
Brief Title: Clinical Study of Customized Adjustable Oral in Treatment of Patients With Obstructive Sleep Apnea Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY-2018-5-10
Record Dates: First submitted 2018-09-24; First posted 2018-11-05 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-09

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: Orthodontic Appliances; Cone-Beam Computed Tomography
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: Twenty-four patients diagnosed with OSAS in different degrees,who cannot tolerate continuous positive air pressure use and reject a surgical approach, were treated with adjustable customized oral appliances and evaluated with cone-beam computed tomography and polysomnography.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with OSAS in different degrees (Experimental): OSAS patients will be treated with an adjustable oral appliance and evaluated with cone-beam computed tomography and polysomnography.
  Interventions: Device: Adjustable Oral Appliance

INTERVENTIONS:
Device: Adjustable Oral Appliance — Adjustable Oral Appliance consist of plastic maxillary occlusal splint，mandible occlusal splint and adjustable connecting rod.It could offer a non-invasive form of treatment but also achieve a good therapeutic effect

SUMMARY:
The oral appliances (OAs) are considered to be an effective treatment modality for snoring and various forms of obstructive sleep apnea syndrome (OSAS). They facilitate the displacement of the mandible anteriorly and widen the upper airway during sleep. Lateral cephalometry has been used for the two-dimensional evaluation of upper airway form with several limits.The purpose of present study is to investigate an accurate three-dimensional (3D) volume analyses with cone beam computed tomography (CBCT) scans to confirm the effects of OAs on the upper airway in patients with OSAS.The investigators aim to enroll twenty-four patients with mild,moderate or severe OSAS, intolerant to continuous positive air pressure therapy and rejection a surgical approach,who will be treated with adjustable customized OAs and evaluated with CBCT and polysomnography. Upper airway form was examined and the volume was measured in two different areas. Specific planes have been considered to match the data and calculate the benefit obtained with therapy.

DETAILED DESCRIPTION:
Obstructive sleep apnea syndrome (OSAS) represents the most common nocturnal respiratory disease characterized by repetitive episodes of partial or complete upper airway collapse or narrowing during sleep,associated with phasic oxygen desaturation.Failure to recognize this condition could lead to an increased risk of cardiovascular diseases, daytime sleepiness, road accidents, a reduced cognitive capacity, with a decline of the quality of life.According to the American Association of Sleep Medicine,the diagnostic standard of the OSAS is the polysomnographic exam, which allows to assess the gravity of OSAS in relation to the Apnea Hypopnea Index (AHI) within an hour:slight (AHI<5), moderate (5<AHI<30) and severe (AHI>30). Epidemiological investigations has shown that the prevalence rate of OSAS is 2-4% of the total population,whereas the percentage of undiagnosed OSAS remains very high with progression to dangerous complications.

OSAS treatment modalities include proper body position, slimming,continuous positive air pressure(CPAP),surgical procedures and oral appliances use. OA are dental devices that improve OSAS by producing a structural change of the upper airways, in order to mechanically increase the pharyngeal diameters, keep the tongue from falling backwards and to stiffen the pharyngeal muscles longitudinally.Recently, OAs is growing more popular due to its superiority in the treatment of the OSAS.It offers a non-invasive form of treatment but also achieve a good therapeutic effect. Traditionally, the effects of functional appliances are evaluated using two-dimensional (2D) radiographs, but the reproducibility of 2D is complex, and overlapping images are difficult to assess. Cone-beam computed tomography (CBCT) provides more accurate and reproducible imaging for assessing all craniofacial skeletal structures.

The objective of this study was to evaluate, in a 6-months follow-up study, the effect of costumed adjustable oral appliance in OSAS patients both through the comparison of the polysomnographic analysis, and also through the volumetric measurements of the pharyngeal airway by using the cone beam computed tomography.

Twenty-four patients,aged 18 to 50 years,in whom the diagnosis of OSAS was made following polysomnography in a sleep laboratory will be enrolled between September 2018 and November 2018.All patients will also undergo a systematic dental examination by a dentist, which put an indication to the use of OA, based also on the craniofacial features assessment. The Epworth Sleepiness Scale (ESS) will be used to evaluate daytime sleepiness.

They then will be fitted with a costumed adjustable oral appliance. The appliances are taken with a mandibular advancement of 2-3 mm and vertical rise of 4-5 mm, that is, the vertical position set at the minimum occlusal elevation to allow mandibular advancement and to avoid backward rotation. The participants were asked to wear the test appliance for 7 nights, and in case of compliance,application it every night at least for 6 months. The selected patients will be record their usage of the appliance and any adverse effects in a treatment journal.

The research focus on the following outcomes: sleep apnea and the the volumetric changes of the upper airway. All patients were radiographically evaluated with a specific diagnostic examination: the cone beam computed tomography scan. For each patient, 3 CBCT scans were performed positioning his head in a neutral way and were performed without swallowing or respiratory movements during inspiration at rest: the first one before the therapy, the second after 3 months and the second after 6 months. Data obtained through CBCT scans have been exported in DICOM format and analyzed with a specific software (MIMICS-Materialise Interactive Medical Image Control System, Leuven, Belgium).The pharyngeal area around the velopharynx and oropharynx has been considered in which the origin of apneas is mainly found.Three planes have been built, an upper, a middle, and lower one, all perpendicular to the median sagittal plane of symmetry to obtain 2 areas, a superior and an inferior one.

ELIGIBILITY:
Inclusion Criteria:

* Apnea-hypopnea index(AHI)between 5/h and 45/h
* Aged between 18 and 50 years old
* Intolerance to continuous positive airway pressure or surgery
* Body Mass Index(BMI) <35kg/m
* Those who are competent to give written informed consent
* Have adequate tooth support to retain the oral appliance

Exclusion Criteria:

* Previous or current treatment for OSAS
* Presence of respiratory/sleep disorders other than obstructive sleep apnea
* Medication usage that could influence respiration or sleep
* Concurrent unstable cardiovascular disease,neurological or mental disorders
* Active periodontal endodontic disease or open bite
* Temporomandibular joint disorders
* Loss of posterior dental support to undermine the retention of oral appliance
* Pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
change in apnea hypopnea index(AHI) | 3,6 and 10 months
  the change from apneas hypopneas per hour of sleep registration of the subjects fitted with oral appliance at 3,6 and 10 months

SECONDARY OUTCOMES:
change in apnea index(AI) | 3,6 and 10 months
  the change from apneas per hour of sleep registration of the subjects fitted with oral appliance at 3,6 and 10 months
change in lowest blood oxygen saturation | 3,6 and 10 months
  the change from the ratio of the content of oxyhaemoglobin to the content of oxygenic hemoglobin in the blood of the subjects at 3,6 and 10 months
change in minimal volume/transverse diameter/sagittal diameter/cross-sectional area of the velopharyngeal segment of the subjects | 3,6 and 10 months
  the change from velopharyngeal segment of upper airway is the region between two planes pass separately through the posterior nasal spine point (PNS) and the tip of soft palate point(U),which are parallel to frankfort horizontal plane(FH) after 3,6 and 10 months
change in minimal volume/transverse diameter/sagittal diameter/cross-sectional area of the oropharyngeal segment of upper airway | 3,6 and 10 months
  the change from oropharyngeal segment of upper airway is the region between two planes pass separately through the highest point of epiglottis(EP) and the tip of soft palate point(U),which are parallel to frankfort horizontal plane(FH) at 3,6 and 10 months

CONTACTS AND LOCATIONS:
Overall Officials: rongjian Lu, doctor, Study Director — Chinese PLA 307 Hospital
Locations (1):
- Chiese PLA 307 hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No